CLINICAL TRIAL: NCT06061367
Title: Influence of Lower Extremity Muscles Strength on Physical Function, Biomechanical Gait Parameters and Reported Outcome After Total Knee Arthroplasty
Brief Title: Muscles Strength and Gait Parameteres After TKA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Professor, Medical University of Warsaw
Other Study IDs: WarsawMU/MUSABGP
Record Dates: First submitted 2023-07-29; First posted 2023-09-29 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Arthritis Knee; Gait Biomechanics; Total Knee Arthroplasty; Muscle Strength; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total Knee Arthroplasty (TKA) is actually the most effective treatment option for patients with end-stage osteoarthritis (OA). However, nearly 20% of patients who underwent TKA remain unsatisfied with their clinical outcome. Investigating modifiable factors that limit knee functioning following TKA we may notice the significance of lower limb muscles strength. Gait pattern is also affected by OA, as arthritic knee joint cannot provide proper range of motion (ROM) and stability.Therefore any deviation in biomechanics should be noticed and analyzed. After TKA patients' physical function may change, but the study should be conducted to prove whether it improves or not. Patient-reported outcome defined by OKS (Oxford Knee Score) and FJS (Forgotten Joint Score) questionnaires will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* III° or IV° grade knee osteoarthritis
* Age over 50
* Patients with signed consent

Exclusion Criteria:

* Undergone total hip replacement
* Previous femur fracture in anamnesis
* Undergone corrective osteotomy
* Active/ Chronic neoplastic disease
* Significant deformation of lower limb axis
* Mental disorders
* Muscular disorders

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 50 years old with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle strength measurement with a use of dynamometer | 6 months
  Analysis of pre- and postoperative strength of lower limb muscles. Assessment of force [N] generated by knee flexors, knee extensors, hip adductors and hip abductors with a use of a hand-held dynamometer.
Gait biomechanics analysis - step length | 6 months
  Analysis of pre- and postoperative parameters of gait pattern and biomechanics with a use of Baiobit device (wearable motion analysis system). Subjected to the analysis will be the step length (in meters).
Gait biomechanics analysis - gait speed | 6 months
  Analysis of pre- and postoperative parameters of gait pattern and biomechanics with a use of Baiobit device (wearable motion analysis system). Subjected to the analysis will be the gait speed (metre per second).
Gait biomechanics analysis - phases of gait | 6 months
  Analysis of pre- and postoperative parameters of gait pattern and biomechanics with a use of Baiobit device (wearable motion analysis system). Subjected to the analysis will be the swing and the stance phase of gait (% of the gait cycle).
Gait biomechanics analysis - step duration | 6 months
  Analysis of pre- and postoperative parameters of gait pattern and biomechanics with a use of Baiobit device (wearable motion analysis system). Subjected to the analysis will be the duration of left and right step (in seconds).
Physical function assessment based on standardized test | 6 months
  Analysis of pre- and postoperative physical function on the basis of Up and Go test.

SECONDARY OUTCOMES:
Patient-reported outcome - Oxford Knee Score | 6 months
  Pre- and postoperative evaluation of Oxford Knee Score. Patients will be asked 12 closed-end questions. 5 possible answers to choose. The scoring system is from 0 to 4 for each answer. Total score ranges from 0 to 48, where 0 is the poorest outcome, and 48 is the best one.
Patient-reported outcome - Forgotten Joint Score | 6 months
  Pre- and postoperative evaluation of Forgotten Joint Score. The questionnaire is based on 12 questions. Total score ranges from 0 to 100. Higher score on the questionnaire, means better results were obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Poland